CLINICAL TRIAL: NCT03341767
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety, Tolerability, Pharmacokinetics and Efficacy of Clofazimine (CFZ) in Cryptosporidiosis
Brief Title: A Phase 2A Evaluation of the Safety, Tolerability, Pharmacokinetics, Efficacy of Clofazimine (CFZ) in Cryptosporidiosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); The Emmes Company, LLC (Industry); Calibr, a division of Scripps Research (Other); Liverpool School of Tropical Medicine (Other); University of Virginia (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other)
Responsible Party: Principal Investigator, Wes Van Voorhis, Professor, School of Medicine, Allergy & Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFZ-001; CC-ID8 (Other: The Emmes Corporation)
Record Dates: First submitted 2017-10-26; First posted 2017-11-14 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Cryptosporidiosis
Keywords: HIV; Cryptosporidium; Clofazimine
MeSH Terms: conditions — Cryptosporidiosis | interventions — Clofazimine

STUDY DESIGN:
Intervention Model Description: Parallel assignment, placebo-controlled with later arm for pharmacokinetics
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clofazimine (Experimental): Subjects >/=50 kg: Clofazimine two 50mg gelatin capsules taken orally every 8 hours for 5 days Subjects <50 kg: Clofazimine 50mg gelatin capsule taken orally every 8 hours for 5 days
  Interventions: Drug: Clofazimine
- Placebo (Placebo Comparator): Placebo gelatin capsule(s) taken orally every 8 hours for 5 days.
  Interventions: Drug: Placebo
- Clofazimine, no diarrhea (Experimental): Subjects >/=50 kg: Clofazimine two 50mg gelatin capsules taken orally every 8 hours for 5 days Subjects <50 kg: Clofazimine 50mg gelatin capsule taken orally every 8 hours for 5 days
  Interventions: Drug: Clofazimine

INTERVENTIONS:
Drug: Clofazimine — 50 or 100 mg micronized Clofazimine suspended in an oil-wax base in a gelatin capsule
  Other Names: Lamprene
  Arms: Clofazimine; Clofazimine, no diarrhea
Drug: Placebo — Oil-wax in gelatin capsule
  Other Names: Placebo (for Clofazimine)
  Arms: Placebo

SUMMARY:
This study evaluates the safety, tolerability, pharmacokinetics, and efficacy of treating Cryptosporidiosis in HIV positive patients with Clofazimine. Half of the HIV positive patients with Cryptosporidiosis enrolled will be treated with Clofazimine while the other half will be given placebo. An additional group of HIV positive patients without Cryptosporidium infection or diarrhea will be given Clofazimine to assess the differences in pharmacokinetics between HIV positive patients with and without Cryptosporidiosis and diarrhea.

DETAILED DESCRIPTION:
Cryptosporidiosium infection and diarrhea is a life-threatening infection in children 6-18 months and in immunocompromised patients. However, Nitazoxanide, the only drug approved for treatment of Cryptosporidiosis, showed little-to-no efficacy in HIV positive patients and low efficacy in malnourished children.

Recently, Love MS et al reported that Clofazimine inhibited proliferation of both Cryptosporidium parvum and C. hominis in vitro and reduced shedding in a mouse model of acute C. parvum infection. Clofazimine has been approved for treatment of leprosy for decades and more recently for the treatment of drug-resistant Mycobacterium tuberculosis. Safety and pharmacokinetics of Clofazimine are well documented for a variety of patient populations, but not for HIV positive patients or patients with diarrhea. Thus, this clinical trial seeks to determine the efficacy of 50 or 100 mg of Clofazimine administered 3 times daily for 5 days on fecal shedding of Cryptosporidium oocysts in HIV positive patients, as well as safety, tolerability, and pharmacokinetics in this patient population.

ELIGIBILITY:
Part A:

Inclusion Criteria:

* Male or Female, Aged 18-65 years old, HIV positive, Cryptosporidium positive by qPCR.
* HIV infection and on stable anti-retroviral therapy treatment for at least 2 weeks
* Weight >78 lbs/35.4 kg
* Presents with diarrhea defined as a condition of three or more loose stools per day that has persisted for 3 days or longer
* If female, either not of reproductive potential (post-menopause, or status-post surgical sterilization) or using highly effective contraception (<1% failure, e.g., intrauterine contraceptive device in place or using injectable contraception) or willing to begin highly effective contraception (probably injectable contraception) and continue for the presumed exposure period of Clofazimine (54 days after initiation of treatment)
* Willing and able to provide signed written informed consent or witnessed oral consent in the case of illiteracy, prior to undertaking any trial-related procedures

Exclusion Criteria:

* Any condition for which participation in the study, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments
* Fever >38.0˚C at presentation
* Subjects will be screened for evidence of active tuberculosis based on sputum production, fever and chest x-ray. Those with sputum production will be tested by Acid Fast Bacilli stain of sputum smear and/or by GeneXpert testing. Those with positive sputum or chest x-ray suggestive of tuberculosis will be excluded from this study and referred for treatment.
* Is critically ill, or in the judgment of the investigator has a prognosis that could lead to imminent mortality within 60 days or compromise participation in the trial or endanger the subject by entering the trial.
* History of allergy or hypersensitivity to Clofazimine.
* Significant cardiac arrhythmia requiring medication.
* Electrocardiogram exclusions based on the means from triplicate electrocardiograms performed on Day -1:

  1. Marked prolongation of QT/QTc interval, e.g., confirmed demonstration of QTcF or QTcB interval >450 ms
  2. Pathological Q waves (defined as >40 ms or depth >0.4 to 0.5mV);
  3. Electrocardiogram evidence of ventricular pre-excitation
  4. Electrocardiogram evidence of complete or incomplete left bundle branch block or right bundle branch block
  5. Electrocardiogram evidence of second or third degree heart block
  6. Intraventricular conduction delay with QRS duration >120 ms
  7. Bradycardia as defined by sinus rate <50 bpm.
* History of additional risk factors for Torsade de Pointes, e.g., heart failure; bradycardia with HR<50 bpm, untreated hypothyroidism, hypokalemia <3.0 mEq/L
* Family history of long QT syndrome
* Use of concomitant medications that markedly prolong the QT/QTc interval or are predicted to have drug-drug interactions with Clofazimine that may lead to toxicity from the partner drug including Amiodarone, Amprenavir, Atazanavir, Bedaquiline, Bepridil, Chloroquine, Chlorpromazine, Cisapride, Clarithromycin, Cyclobenzaprine, Darunavir, Delamanid, Disopyramide Dofetilide, Domperidone, Droperidol, Erythromycin, Fosamprenavir, Halofantrine, Haloperidol, Ibutilide, Indinavir, Levomethadyl, Lopinavir, Mesoridazine, Methadone, Nelfinavir, Pentamidine, Pimozide, Procainamide, Quinidine, Ritonavir, Simiprinivir, Sotalol, Sparfloxacin, Thioridazine, or Tiprinivir
* Pregnant and lactating women (screening pregnancy test for females and pregnancy test at the discharge follow up visit)
* Use of systemic corticosteroids or anti-cryptosporidial treatments within the 28 days preceding Day -1
* Subjects with clinically significant laboratory value abnormalities at screening including but not limited to (note: exclusionary results may not be returned until after enrollment but should be confirmed by the time of the beginning of administration of study drug):

  1. Hemoglobin <5 g/dL
  2. Serum potassium <3.0 mEq/L
  3. Aspartate Aminotransferase or Alanine Aminotransferase ≥3.0 x ULN

Part B:

Same Eligibility Criteria except without diarrhea and is Cryptosporidium negative by qPCR.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Reduction in Cryptosporidium fecal shedding following Clofazimine administration | 5 days
  The reduction in the (log) number of Cryptosporidium shed in stools in the first collected stool of the day over a 6-day period and compared to placebo recipients, as measured by quantitative polymerase chain reaction (qPCR) in stool samples and analyzed by a mixed effect ANCOVA analysis in subjects treated according to protocol (ATP).
Pharmacokinetics (area under curve) of Clofazimine in HIV-infected subjects with Cryptosporidium and diarrhea versus HIV-infected subjects without Cryptosporidium infection or diarrhea | 5 days
  Clofazimine in plasma will be assessed via area under curve.
Peak plasma concentration of Clofazimine in HIV-infected subjects with Cryptosporidium and diarrhea versus HIV-infected subjects without Cryptosporidium infection or diarrhea | 5 days
  Clofazimine in plasma will be assessed via Cmax and time to reach Cmax (Tmax).
Pharmacokinetics (Ke) of Clofazimine in HIV-infected subjects with Cryptosporidium and diarrhea versus HIV-infected subjects without Cryptosporidium infection or diarrhea | 5 days
  Clofazimine in plasma will be assessed via Ke determined after the last dose on day 5.
Stool pharmacokinetics of Clofazimine in HIV-infected subjects with Cryptosporidium and diarrhea versus HIV-infected subjects without Cryptosporidium infection or diarrhea | 5 days
  The total daily amount of CFZ eliminated in stool will be assessed on Study Day 2 (2nd dose day), Study Day 5 (last dose day), and Study Day 6 (concentration of CFZ in stool before discharge).
Frequency and severity of solicited adverse events (AEs) | 5 days
  Frequency and severity of solicited AEs throughout study product administration
Frequency, severity, and relationship to study product of unsolicited AEs | 55 days
  Frequency, severity, and relationship to study product of unsolicited AEs throughout the course of the study
Occurrence of serious adverse events (SAEs), suspected unexpected serious adverse reactions (SUSARs), and adverse events of special interest (AESI). | 55 days
  Occurrence of SAEs, SUSARs, and AESIs throughout the course of the study. AESI include: QT prolongation measured via 12-lead electrocardiogram, liver toxicity, skin discoloration and other skin related AEs/abnormalities (subjects will be evaluated for discoloration of skin of the palms and of the sclera and oral mucous membranes), GI-related AEs.

SECONDARY OUTCOMES:
Evaluation of time to negative ELISA signal in subjects randomized to Clofazimine versus placebo | 6 days
  Evaluate days required to test negative for Cryptosporidium by ELISA test in subjects randomized to Clofazimine versus placebo.
Characterization of the reduction in the number of diarrheal episodes following administration of CFZ relative to placebo. | 6 days
  To characterize the reduction in the number of diarrheal episodes following administration of CFZ relative to placebo.
Characterization of the stool volume following administration of CFZ relative to placebo. | 6 days
  To characterize the stool volume following administration of CFZ relative to placebo.
Characterization of the stool consistency following administration of CFZ relative to placebo. | 6 days
  To characterize the stool consistency based on a defined diarrheal stool grading scale following administration of CFZ relative to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Wes Van Voorhis, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme (MLW), Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Love MS, Beasley FC, Jumani RS, Wright TM, Chatterjee AK, Huston CD, Schultz PG, McNamara CW. A high-throughput phenotypic screen identifies clofazimine as a potential treatment for cryptosporidiosis. PLoS Negl Trop Dis. 2017 Feb 3;11(2):e0005373. doi: 10.1371/journal.pntd.0005373. eCollection 2017 Feb. PMID 28158186
- [Derived] Zhang CX, Love MS, McNamara CW, Chi V, Woods AK, Joseph S, Schaefer DA, Betzer DP, Riggs MW, Iroh Tam PY, Van Voorhis WC, Arnold SLM. Pharmacokinetics and Pharmacodynamics of Clofazimine for Treatment of Cryptosporidiosis. Antimicrob Agents Chemother. 2022 Jan 18;66(1):e0156021. doi: 10.1128/AAC.01560-21. Epub 2021 Nov 8. PMID 34748385
- [Derived] Iroh Tam P, Arnold SLM, Barrett LK, Chen CR, Conrad TM, Douglas E, Gordon MA, Hebert D, Henrion M, Hermann D, Hollingsworth B, Houpt E, Jere KC, Lindblad R, Love MS, Makhaza L, McNamara CW, Nedi W, Nyirenda J, Operario DJ, Phulusa J, Quinnan GV, Sawyer LA, Thole H, Toto N, Winter A, Van Voorhis WC. Clofazimine for Treatment of Cryptosporidiosis in Human Immunodeficiency Virus Infected Adults: An Experimental Medicine, Randomized, Double-blind, Placebo-controlled Phase 2a Trial. Clin Infect Dis. 2021 Jul 15;73(2):183-191. doi: 10.1093/cid/ciaa421. PMID 32277809
- [Derived] Nachipo P, Hermann D, Quinnan G, Gordon MA, Van Voorhis WC, Iroh Tam PY. Evaluating the safety, tolerability, pharmacokinetics and efficacy of clofazimine in cryptosporidiosis (CRYPTOFAZ): study protocol for a randomized controlled trial. Trials. 2018 Aug 23;19(1):456. doi: 10.1186/s13063-018-2846-6. PMID 30139372